CLINICAL TRIAL: NCT00789139
Title: Recurrence of Arrhythmias After Pulmonary Veins Isolation Detected by ICM
Acronym: RAPID XT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr Ange FERRACCI (Other)
Responsible Party: Sponsor-Investigator, Dr Ange FERRACCI, CARDIOLOGIST, Hospital St. Joseph, Marseille, France
Organization: Hospital St. Joseph, Marseille, France (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RAPIDXT
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AF monitoring by ICM (Other): Only one arm
  Interventions: Device: ICM Implantation

INTERVENTIONS:
Device: ICM Implantation — Sub cutaneous implantation of the ICM

SUMMARY:
Post Marketing study, Interventional, Prospective, non randomised

Describe how the MD is using the information of the ICM in addition of standard FU(clinical exam and holter 24h)post AF ablation(1 year FU).

ELIGIBILITY:
Inclusion Criteria:

* AF thermoablation indication
* Informed Consent signed,
* Age between 18 & 75

Exclusion Criteria:

* Participation to other clinical trial
* Non compliant patient
* Pregnant women
* Left Atrial thrombus
* Endocarditis, infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-10; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Clinical exam and ECG record | one month, 3 months, 6 months , 12 months

CONTACTS AND LOCATIONS:
Overall Officials: ANGE FERRACCI, md, Principal Investigator — Unity Health Toronto; ANDRE PISAPIA, MD, Study Director — Unity Health Toronto
Locations (1):
- Saint Joseph Hospital, Marseille, France